CLINICAL TRIAL: NCT06489197
Title: Ivonescimab(AK112) Combined With Chemotherapy as the First-line Treatment in Patients With Advanced Esophageal Squamous Cell Carcinoma (ESCC): A Single Arm , Phase II Trial
Brief Title: AK112 Combined With Chemotherapy as the First-line Treatment in Advanced Esophageal Squamous Cell Carcinoma Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK112-IIT-009
Record Dates: First submitted 2024-06-28; First posted 2024-07-05 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-06

CONDITIONS: ESCC; Advanced Esophageal Squamous Cell Carcinoma
MeSH Terms: interventions — Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): Ivonescimab combined with albumin paclitaxel and cisplatin
  Interventions: Drug: Ivonescimab combined with albumin paclitaxel and cisplatin

INTERVENTIONS:
Drug: Ivonescimab combined with albumin paclitaxel and cisplatin — Ivonescimab (20mg/kg, intravenous infusion, d1, Q3W) combined with albumin paclitaxel (220mg/m2, intravenous infusion, d1, Q3W) and cisplatin (75mg/m2, intravenous infusion, d1, Q3W), of which the maximum treatment time of chemotherapy was up to six cycles, and the maximum treatment time of AK112 was 24 months.

SUMMARY:
This is a single arm，phase 2 study evaluating the safety and efficacy of Ivonescimab(AK112) combined with chemotherapy in the treatment of advanced esophageal squamous cell carcinoma (ESCC). In this study, patients with advanced esophageal squamous cell carcinoma who had not received any systematic treatment in the past will be enrolled.

The research will be conducted in two stages. In the first part, 6 patients were enrolled in the group. After the last subject in the group completed at least 21 days of observation after the first medication, the researchers will conduct a preliminary safety and effectiveness assessment. If the safety and tolerability are good, it will enter the second expansion part till the study enrolled 30 patients. Patients who met the inclusion criteria were treated with AK112 (20mg/kg, intravenous infusion, d1, Q3W) in combination with albumin paclitaxel (220mg/m2, intravenous infusion, d1, Q3W) and cisplatin (75mg/m2, intravenous infusion, d1, Q3W), of which the maximum treatment time of chemotherapy was up to six cycles, and the maximum treatment time of AK112 was 24 months. Patients received regular and periodic reviews, with imaging evaluations every 6 weeks.

DETAILED DESCRIPTION:
Part 1: Safety introduction phase, evaluate the safety and tolerability of AK112 combined with chemotherapy (albumin paclitaxel and cisplatin). Plan to enroll 6 advanced ESCC subjects who have not undergone any systematic anti-tumor treatment in the past. After completing at least 21 days of observation after the first medication of the last enrolled subject, the researchers will conduct preliminary safety and efficacy evaluations. If the safety and tolerability are good, and preliminary therapeutic signals are observed, it will enter the stage of expansion into the group. Researchers may also discuss adjusting the AK112 dose, albumin paclitaxel dose, or cisplatin dose based on the specific situation during the DLT observation period, and then enroll new subjects for the safety introduction phase evaluation of the treatment plan in the study group.

DLT definition: Within 21 days after the first administration, the subject experiences the following drug-related toxic reactions (according to NCI CTC AE 5.0 toxicity evaluation criteria): hematological toxicity level 4 or above or non hematological toxicity level 3 or above (excluding hair loss).

Part 2: Expand the enrollment stage, to further evaluate the efficacy and safety of AK112 combined with albumin paclitaxel and cisplatin in first-line treatment of advanced ESCC. During the expansion phase, 30 subjects will be enrolled, and a comprehensive discussion will be conducted based on the safety and efficacy data from the safety introduction phase to determine the dosage.

ELIGIBILITY:
Inclusion Criteria:

1. Signed the informed consent；
2. Male or female patients ≥18 and ≤ 75 years old;
3. ECOG physical status score is 0 or 1;
4. Patients with non resectable or metastatic advanced ESCC confirmed by pathological ocytological examination;
5. No previous systemic treatment;
6. Expected survival time ≥ 3 months;
7. Patients must have at least one measurable metastatic lesion according to RECIST version 1.1;
8. Normal organ function:

   1. Hematology :Absolute neutrophil count (ANC) ≥ 1.5 × 109/L (1500/mm3); Platelet count ≥ 100 × 109/L (100000/mm3); Hemoglobin ≥ 90g/L;
   2. Kidney:The calculated value of creatinine clearance rate (CrCl) is ≥ 50 mL/min;Normal urine routine, urine protein<2+or 24-hour (h) urine protein quantification<1.0 g;
   3. Liver:Total serum bilirubin (TBiL) ≤ 1.5 × ULN;AST and ALT ≤ 2.5 × ULN; For subjects with liver metastasis, AST and ALT can be ≤ 5 × ULN;Serum albumin (ALB) ≥ 30g/L;
   4. Normal coagulation function, international standardized ratio (INR) ≤ 1.5 x ULN, prothrombin time (PT) and activated partial thromboplastin time (APTT) ≤ 1.5 x ULN;
9. Women of childbearing age must undergo a pregnancy test (serum or urine) with a negative result within 14 days before enrollment, and voluntarily use appropriate methods of contraception during the observation period and within 8 weeks after the last administration of the study drug; For males, surgical sterilization or agreement to use appropriate methods of contraception during observation and within 8 weeks after the last administration of study medication should be considered;
10. Comply with the scheduled visits, treatment plans, laboratory tests, and other requirements of the study;

Exclusion Criteria:

1. Local advanced esophageal squamous cell carcinoma that can be curative through surgery or potentially cured through radiation therapy;
2. Suffering from other malignant tumors within the 5 years prior to enrollment. Patients with other malignant tumors that have been cured by local treatment, such as basal or cutaneous squamous cell carcinoma, superficial bladder cancer, cervical or breast cancer in situ, are not excluded;
3. Active bleeding signs of the lesion are displayed under endoscopy;
4. Currently participating in intervention clinical research treatment, or having received other research drugs or used research instruments within 4 weeks before the first administration;
5. Receiving immunotherapy in the past, including immune checkpoint inhibitors (such as anti-PD-1/L1 antibodies, anti-CTLA-4 antibodies, anti-TIGIT antibodies, anti-LAG3 antibodies, etc.), immune checkpoint agonists (such as ICOS, CD40, CD137, GITR, OX40 antibodies, etc.), immune cell therapy, or any other treatment targeting the immune mechanism of tumors;
6. Received systemic non-specific immunomodulatory therapy (such as interleukin, interferon, thymosin, etc.) within 2 weeks before the first administration;
7. Active autoimmune diseases that require systemic treatment (such as the use of disease relieving drugs, glucocorticoids, or immunosuppressants) have occurred within 2 years prior to the first administration.
8. The study is currently undergoing systemic glucocorticoid therapy (excluding local glucocorticoids through nasal spray, inhalation, or other routes) or any other form of immunosuppressive therapy within 7 days prior to the first administration; Note: Physiological doses of glucocorticoids (≤ 10 mg/day of prednisone or equivalent) are allowed to be used;
9. Clinically significant gastrointestinal obstruction, gastrointestinal perforation, intra-abdominal abscess, fistula formation, etc. occur within 6 months before the first administration;
10. Active, uncontrolled, or recurrent inflammatory gastrointestinal diseases (such as Crohn's disease, ulcerative colitis, radiation enteritis, hemorrhagic enteritis, chronic diarrhea, etc.);
11. Previous history of myocarditis, cardiomyopathy, and malignant arrhythmia. Unstable angina, myocardial infarction, congestive heart failure (classified as grade 2 or above according to the New York Heart Association functional classification) or vascular disease (such as aortic aneurysm with a risk of rupture) that requires hospitalization within 12 months prior to the first administration, or other cardiac damage that may affect the safety evaluation of the investigational drug (such as poorly controlled arrhythmias, myocardial ischemia);
12. Any arterial thromboembolism events, NCI CTCAE 5.0 grade 3 or above venous thromboembolism events, transient ischemic attacks, cerebrovascular accidents, hypertensive crises, or hypertensive encephalopathy occurred within 6 months prior to the first administration; Currently, there is hypertension and after treatment with oral antihypertensive drugs, the systolic blood pressure is ≥ 160mmHg or the diastolic blood pressure is ≥ 100mmHg;
13. Severe infections occurring within 4 weeks prior to the first administration, including but not limited to comorbidities requiring hospitalization, sepsis, or severe pneumonia; Active infections that have received systemic anti infective treatment within 2 weeks prior to the first administration (excluding antiviral treatment for hepatitis B or C);
14. Subjects with active hepatitis B are required to receive anti hepatitis B virus treatment during the study treatment; Active hepatitis C subjects (HCV antibody positive and HCV RNA levels above the detection limit);
15. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation;
16. If the toxicity of previous anti-tumor treatments has not improved, it is defined as the toxicity has not returned to level 0 or 1 of NCI CTCAE 5.0, or the level specified in the inclusion/exclusion criteria, except for hair loss;
17. Known to be allergic to any component of any investigational drug; Known medical history of severe hypersensitivity reactions to other monoclonal antibodies;
18. If a live vaccine or attenuated live vaccine is administered within 30 days prior to the first administration, or if a live vaccine or attenuated live vaccine is planned to be administered during the study period, the use of inactivated vaccines is allowed;
19. Known history of mental illness, drug abuse, alcohol or drug abuse;
20. Pregnant or lactating women;
21. Those who have undergone major surgical procedures or experienced severe trauma within 30 days prior to the first administration, or those who have planned major surgical procedures within 30 days after the first administration (as determined by the investigator); Minor local surgeries were performed within 3 days prior to the first administration (excluding peripheral venous puncture, central venous catheterization, and intravenous infusion port implantation);
22. During the screening period, imaging showed significant necrosis and cavities in the tumor, and the researchers determined that entering the study would pose a risk of bleeding; Tumors invade important blood vessels and organs; Tumor mediastinal lymph node metastasis invading the trachea, main bronchus, or at risk of developing esophagotracheal fistula or esophagopleural fistula;
23. Have a history of severe bleeding tendency or coagulation dysfunction; There are significant clinically significant bleeding symptoms within one month prior to the first administration; Patients who have previously or currently require long-term therapeutic anticoagulation therapy (such as atrial fibrillation patients who meet CHADS2 score ≥ 2);
24. The researcher believes that there are other potential risks that are not suitable for participation in this study;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-16 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate,ORR | 6 months
  Defined as the proportion of patients who achieved complete response (CR) and partial response (PR) according to RECIST v1.1.

SECONDARY OUTCOMES:
Overall survival,OS | 24 months
  Defined as the time between signing the informed consent form to death due to various causes.
Progression free Survival,PFS | 12 months
  Defined as the time between signing the informed consent form to the disease progression (according to RECIST v1.1 criteria) or death due to any cause.
Disease Control Rate,DCR | 6 months
  Defined as the proportion of patients who achieved complete response (CR), partial response (PR), and stable disease (SD) according to RECIST v1.1.
Duration of Response,DoR | 6 months
  Defined as the time from response(when CR or PR is first diagnosed) to disease progression or death due to any cause.

OTHER OUTCOMES:
Incidence of adverse events | 24 months
  Use NCI-CTCAE version 5.0 for classification and grading.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No